CLINICAL TRIAL: NCT02255617
Title: A Prospective, Single Center, Open Label Trial of Fecal Microbiota Transplantation (FMT) in the Management of Hepatic Encephalopathy (HE): a Pilot Study
Brief Title: Fecal Microbiota Transplantation (FMT) in the Management of Hepatic Encephalopathy (HE): a Pilot Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Dina Kao, Assistant Professor, University of Alberta
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 47057
Record Dates: First submitted 2014-08-26; First posted 2014-10-02 (Estimated); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Hepatic Encephalopathy
MeSH Terms: conditions — Hepatic Encephalopathy | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fecal Microbiota Transplant (Experimental): Single arm open label FMT administered at Week 0 by colonoscopy and at Weeks 1-4 by enema
  Interventions: Biological: Fecal Microbiota Transplant

INTERVENTIONS:
Biological: Fecal Microbiota Transplant — Fecal transplant processed from routinely screened universal donors

SUMMARY:
The purpose of this study is to determine if FMT can reverse Hepatic Encephlopathy (HE) in cirrhotic patients who continue to have breakthrough episodes of HE despite maintenance therapy with lactulose and/or rifaximin or metronidazole.

DETAILED DESCRIPTION:
Subjects receive FMT from a single donor by colonoscopy at Week 0 and by enema at Weeks 1-4. HE is measured by Inhibitory Control Test and Stroop as well as serum ammonia levels.

ELIGIBILITY:
Inclusion Criteria:

1. adult (age > 18 years of age) cirrhotic patients of various etiology, on lactulose and/or rifaximin or flagyl for at least 4 weeks as secondary prophylaxis
2. abnormal inhibitory control test, defined as greater than 5 lures.
3. an infectious etiology which may cause HE has been ruled out

Exclusion Criteria:

1. those with tense ascites
2. those who do not provide assent
3. those who are judged to have a life expectancy of less than 3 months,
4. those who had TIPS within 3 months,
5. those with neurologic diseases such as dementia, Parkinson's disease, and structural brain lesions
6. pregnancy
7. those with intestinal obstruction
8. those with alcoholic hepatitis
9. those with active alcohol or substance abuse
10. those without stable social support
11. those who have a concurrent infection, such as SBP, pneumonia or UTI
12. those with creatinine clearance less than 50% compared to baseline
13. those with recent hospital admission, defined as within one month of enrollment, for hepatic encephalopathy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-07-23 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2019-09-23 (Actual)

PRIMARY OUTCOMES:
Portion of participants with normailzation of ICT or Stroop Test during the study | 8 weeks

SECONDARY OUTCOMES:
Proportion of patients with normalization ICT or Stroop test scores at 1 week, 2 weeks, 4 weeks and 8 | 8 weeks
Changes in serum ammonia level pre and post FMT | 8 weeks
Changes in Quality of Life measured by Chronic Liver Disease Questionnaire (CDLQ) pre and post FMT | 8 weeks
Changes in Intestinal Microbiota pre and post FMT | 8 weeks
Serious Adverse Events | 8 weeks
  All serious adverse events up to and including week 8. A serious adverse event is any event which results in any of the following:
  i) Death ii) Colonic perforation iii) Proven infections as defined by the presence of i) spontaneous bacteremia: positive blood cultures in the absence of any other potential source of infection; ii) spontaneous bacterial peritonitis: ascetic fluid PMN equal to or greater than 250/mm3; iii) UTI: urinary leukocyte count greater than 15 cells per HPF and positive urine culture; vi) other infections identified by clinical, radiologic and bacteriologic results.
  iv) Possible infections as defined by i) fever (temp > 37.80 C), ii) leukocytosis (>15,000 mm3) or increased immature neutrophils in blood (>500 mm3), negative cultures and no other signs of infection.
Changes in stool bile acids composition pre and post FMT | 8 Weeks
Changes in stool short chain fatty acids pre and post FMT | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada